CLINICAL TRIAL: NCT01247519
Title: The Effects of Post-hospitalization Telehealth Care in the Patients Who Admitted Via Emergency Department
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chin-Chung Shu, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 200912023R
Record Dates: First submitted 2010-10-05; First posted 2010-11-24 (Estimated); Last update posted 2010-11-24 (Estimated); Status verified 2010-10

CONDITIONS: General Medical Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- observation (No Intervention)
- Intervention (Experimental)
  Interventions: Other: Post-hospitalization care

INTERVENTIONS:
Other: Post-hospitalization care — Post-hospitalization care included telephone call contact for caring after discharge, for opening for question, and for health education.
  Arms: Intervention

SUMMARY:
The investigators will perform and evaluate a post-hospitalization telecare system for compensating the discontinuity from the hospitalist care system.

DETAILED DESCRIPTION:
At present, Taiwan's population has become an aging society since recent decade. Those older than 65 years had achieved 10.4% in 2008. Meanwhile, the proportion of hosts with underlying comorbid illness or immunocomprised status is increasing worldwide. In the trend of aging population, telehealth care will be important to extend the care system in post-hospitalization home care. In the past, thelehealth care has shown a good executive performance in the patients with congestive heart failure and post-operation follow-up. However, in dealing the patients with acute illness needing hospitalization, the telehealth system has not implemented yet. In regard to National health insurance (NHI) of Taiwan, hospitalization costs a lot in overall budget. Reduction of re-hospitalization in those with/without co-morbidity is a important issue for Taiwan NHI. Therefore, we plan to conduct the telehealth care system in post-hospitalization course in those admitted from emergency department. We observe the re-hospitalization rate and analyze the risk factors. In addition, we hypothesize the telehealth care will decrease the rate of re-hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Discharged alive from our hospitalist-care ward to home care
* Match diagnosis of general medicine

Exclusion Criteria:

* Younger than 18 years
* Discharged to care facility other than home
* Died in hospital
* Communication deficits
* No telephone at home
* Patient or family refused

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
readmission | within 30 days after discharge

SECONDARY OUTCOMES:
vist of emergency department | within 30 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan